CLINICAL TRIAL: NCT00005255
Title: Ischemic Heart Disease Incidence and Indices of Body-fat Distribution
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1137; R01HL040844 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia; Obesity

SUMMARY:
To determine the association between ischemic heart disease incidence and anthropometric indices of body-fat distribution.

DETAILED DESCRIPTION:
BACKGROUND:

Previous studies have demonstrated that abdominal obesity can be predictive of ischemic heart disease. These prospective cohort studies employed simple indices of body-fat distribution such as waist-to-hip circumference ratio or subscapular skinfold. Their similar results suggested that increased abdominal obesity conferred a two-fold increased risk of ischemic heart disease among middle-aged men. The two proposed studies permitted testing of alternative fat-distribution indices which might be stronger risk factors for ischemic heart disease incidence than the waist-to-hip-ratio or the subscapular skinfold.

DESIGN NARRATIVE:

Two parallel case-control studies were conducted. In both studies, subjects were measured for girth, skinfold, abdominal sagittal diameter, height, and weight. Analyses for both protocols considered men and women separately. Possible confounders of the association between fat-distribution indices and ischemic heart disease were considered and if required, adjusted for in multivariate analyses. Possible confounders included race, age, tobacco use, alcohol use, diabetes, social class, hypertension, cholesterol levels, and physical activity levels.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-05; Study Completion 1995-04 (Actual)

REFERENCES:
- [Background] Kahn HS, Williamson DF. Abdominal obesity and mortality risk among men in nineteenth-century North America. Int J Obes Relat Metab Disord. 1994 Oct;18(10):686-91. PMID 7866464
- [Background] Kahn HS. Choosing an index for abdominal obesity: an opportunity for epidemiologic clarification. J Clin Epidemiol. 1993 May;46(5):491-4. doi: 10.1016/0895-4356(93)90027-x. PMID 8369048
- [Background] Kahn HS, Simoes EJ, Koponen M, Hanzlick R. The abdominal diameter index and sudden coronary death in men. Am J Cardiol. 1996 Oct 15;78(8):961-4. doi: 10.1016/s0002-9149(96)00479-1. PMID 8888678
- [Background] Kahn HS. The accumulation of visceral adipose tissue may be influenced by intra-abdominal temperature. Obes Res. 1996 May;4(3):297-9. doi: 10.1002/j.1550-8528.1996.tb00550.x. PMID 8732966
- [Background] Kahn HS, Austin H, Williamson DF, Arensberg D. Simple anthropometric indices associated with ischemic heart disease. J Clin Epidemiol. 1996 Sep;49(9):1017-24. doi: 10.1016/0895-4356(96)00113-8. PMID 8780611